CLINICAL TRIAL: NCT06879769
Title: Optimization of Patient Preparation and Imaging Techniques for Cardiac CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Svensson-Marcial, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCTA_2021
Record Dates: First submitted 2025-02-28; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Coronary Computed Tomography Angiography; Contrast Media; Cardiac Output
Keywords: Music intervention; Cardiac Output; CCTA; Beta blockers; Metoprolol
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of Care Group (No Intervention): The participant will receive Seloken orally and Metoprolol I.V. according to the standard of care, with a 1-hour waiting period prior to the examination. Standard of care includes up to 100 mg of oral beta-blockers, with additional intravenous beta-blockers administered if necessary.
- Metoprolol I.V. (Active Comparator): The participant arrives directly at the CT lab without waiting and receives intravenous Metoprolol (up to 15 mg) if systolic blood pressure remains above 105 mmHg and heart rate is over 60 bpm.
  Interventions: Other: Metoprolol I.V.
- Metoprolol I.V. plus 1 hour waiting. (Active Comparator): Participant sits 1 hour in the waiting room and then receives intravenously administered Metoprolol I.V. in the examination room.
  Interventions: Other: Metoprolol I.V. and 1 hour waiting.
- Standard of Care and Music Intervention (Active Comparator): The participant will receive Seloken (Metoprolol) according to clinical routine (up to 100 mg). The participant will also receive noise-canceling headphones and an iPad (or their own device) to select calming music and listen to it one hour before and during the CT scan.
  Interventions: Other: Music Intervention, Seloken (Recordati) orally and Metoprolol I.V.

INTERVENTIONS:
Other: Metoprolol I.V. — The participant will receive intravenous Metoprolol (up to 15 mg) during the CT examination, administered directly at the CT table prior to CCTA.
  Arms: Metoprolol I.V.
Other: Metoprolol I.V. and 1 hour waiting. — The Participant will rest in the waiting room for 1h and then receive intravenous Metoprolol, up to 15 mg.
  Arms: Metoprolol I.V. plus 1 hour waiting.
Other: Music Intervention, Seloken (Recordati) orally and Metoprolol I.V. — The participant will receive Seloken (Metoprolol) according to clinical routine (up to 100 mg) and Metoprolol I.V. (up to 15 mg). The participant will also receive noise-canceling headphones and an iPad (or their own device) to select calming music and listen to it one hour before and during the CT scan.
  Arms: Standard of Care and Music Intervention

SUMMARY:
The goal of this clinical trial is to compare four different methods of reducing heart rate before cardiac imaging. The diagnostic imaging technique used in this study is called Computed Tomography (CT) of the coronary vessels (CCTA). Globally, approximately one-third of patients experience heart-related conditions. Because the heart is a moving organ, imaging presents challenges. A higher heart rate requires increased scanning power, which results in more images and, in some cases, higher radiation exposure that may be harmful. To address this issue, beta-blocker medication is administered before the examination to lower the heart rate. This medication can be given orally, intravenously, or both. While this approach is effective, the most optimal method remains uncertain.

The objectives of this study are:

* To determine whether oral administration of beta-blockers is as effective as intravenous administration in maintaining a stable heart rate during CT imaging.
* To assess whether listening to music during the procedure improves patient comfort and overall experience.

Participants will:

* Be randomly assigned to one of four groups:
* One group will receive beta-blocker medication orally.
* Another group will receive beta-blocker medication intravenously.
* One group will listen to music during the procedure. Participants will report their sensations and experiences before, during, and after the examination.

The study investigators will compare the effectiveness of oral and intravenous beta-blockers, as well as the impact of music, in terms of:

* Heart rate stability and reduction.
* Participant-reported comfort and overall experience.

DETAILED DESCRIPTION:
CT scans are widely utilized due to technological advancements that enable rapid imaging of large anatomical areas, aiding in the assessment of critically ill patients. CT imaging works by detecting how different tissues absorb X-ray radiation, with denser tissues absorbing more. Contrast agents enhance tissue differentiation, but their administration must be carefully managed to minimize potential side effects, such as arrhythmias or kidney impairment.

For CCTA, maintaining a low and stable heart rate is essential to reduce motion artifacts. Beta-blockers are commonly used for this purpose. This study evaluates different patient preparation strategies by comparing the effects of oral and intravenous beta-blockers on heart rate. A total of 240 participants will be enrolled and randomized into four groups, with one group also receiving an auditory intervention involving music.

Heart rate measurements will be obtained using a cardiac output meter, while participants will evaluate their sensory experiences and warmth perception using visual analog scales. The study also aims to determine the optimal timing (s) for imaging following contrast administration, using cardiac output (L/min) and other participant variabels.

A total of 240 participants (120 men and 120 women) will be enrolled and randomized into four groups of 60 individuals per group.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a preexisting referral for a Cardiac CT examination
* Age 18 years or older

Exclusion Criteria:

* Age under 18 years
* Atrial fibrillation
* Pacemaker
* Participation in clinical drug trials
* Contraindications to beta-blockers
* Severe medical conditions
* Challenges in comprehending study information
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | From enrollment to the end of examination, approximately1,5 hours.
  How the heart rate (HR) is impacted by the interventions and the diagnostic images, radiation dose.

SECONDARY OUTCOMES:
Participant anxiety | From enrollment to the end of the examination, approximately 1,5 hours.
  The Visual Analog Scale for Anxiety (VAS-A) is a self-reported scale ranging from 0 to 100, where 0 indicates no anxiety and 100 represents the worst imaginable anxiety.

OTHER OUTCOMES:
Cardiac Output (L/min) | From enrollment to the end of the examination, approximately 1,5 hours.
  Cardiac Output (L/min) is measured before, during and after the Coronary Computed Tomography Angiography (CCTA). Cardiac Output is measured with an Electrical Cardiometry™ (EC) (Aesculon mini; Osypka Medical, Berlin, Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Anders Svensson-Marcial, PhD, Principal Investigator — Karolinska University Hospital, Department of Clinical Science, Intervention and Technology
Locations (1):
- ME Radiologi Huddinge, Karolinska University Hospital, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No
To protect participant data.